CLINICAL TRIAL: NCT00350415
Title: A Double-blind, Randomized, 6-week, Parallel-group Design Clinical Trial to Assess the Safety and Efficacy of Asacol 4.8 g/Day Versus Asacol 2.4 g/Day for the Treatment of Moderately Active Ulcerative Colitis.
Brief Title: A Double Blind Study for the Treatment of Acute Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006444; NCT00336440 (obsolete NCT alias)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis, inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Asacol 2.4 g/day (400 mg tablet)
  Interventions: Drug: Mesalamine
- 2 (Active Comparator): Asacol 4,8 g/day (800 mg tablet), oral, for 6 weeks
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Mesalamine — Asacol 400g/day (400 mg tablet), oral, for 6 weeks
  OR
  Asacol 4,8 g/day (800 mg table), oral, for 6 weeks

SUMMARY:
A Double-blind, Randomized, 6-week, Parallel-group Design Clinical trial to assess the Safety and Efficacy of Asacol 4.8 g/day (800 mg mesalamine tablet) versus Asacol 2.4 g/day (400 mg mesalamine tablet) for the Treatment of Moderately Active Ulcerative Colitis (ASCEND III).

DETAILED DESCRIPTION:
This is a double-blind, randomized, multi-center, multi-national, active-control study in patients who are experiencing a moderately active flare of UC. Patients will be randomly assigned to receive either Asacol 2.4 g/day (400 mg tablet) or Asacol 4.8 g/day (800 mg tablet) for 6 weeks. Patients will be randomized to one of the 2 treatment groups in a 1:1 ratio. The objective of the study is to evaluate the safety and efficacy of Asacol 4.8 g/day (800 mg tablet) compared to Asacol 2.4 g/day (400 mg tablet) in this patient population. Following successful screening, patients will be randomized to one of the two treatment arms. Patients will be evaluated after 6 weeks of treatment with an interim visit after 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-75 years with a confirmed diagnosis of moderately active flare of ulcerative colitis.
* Female patients need to be postmenopausal or using adequate contraception.

Exclusion Criteria:

* Patients with isolated proctitis
* Patients with comorbidities or an investigative or commercialized treatments confounding interpretation of study results or compromising patients' safety in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients (ITT) in each treatment group who achieve treatment success, defined as symptomatic and endoscopic improvement from baseline at Week 6. | Week 6

SECONDARY OUTCOMES:
Proportion of patients (ITT) in pre-defined subgroups in each treatment group who achieve treatment success, defined as symptomatic and endoscopic improvement from baseline at Week 6 and Week 3. | week 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Krzeski, MD, Study Director — Procter and Gamble
Locations (133):
- United States (77):
  - Research Facility, Alabaster, Alabama
  - Research Facility, Birmingham, Alabama
  - Research Facility, Tucson, Arizona
  - Research Facility, Fayetteville, Arkansas
  - Research Facility, Little Rock, Arkansas
  - Research Facility, Anaheim, California
  - Research Facility, Burbank, California
  - Research Facility, Encinitas, California
  - Research Facility, Los Angeles, California
  - Research Facility, Mission Hills, California
  - Research Facility, Orange, California
  - Research Facility, Pasadena, California
  - Research Facility, Roseville, California
  - Research Facility, Sacramento, California
  - Research Facility, San Carlos, California
  - Research Facility, San Francisco, California
  - Research Facility, Lakewood, Colorado
  - Research Facility, Littleton, Colorado
  - Research Facility, Hamden, Connecticut
  - Research Facility, DeLand, Florida
  - Research Facility, Harbor Village, Florida
  - Research Facility, Hollywood, Florida
  - Research Facility, Jacksonville, Florida
  - Research Facility, Panama City, Florida
  - Research Facility, Zephyrhills, Florida
  - Research Facility, Atlanta, Georgia
  - Research Facility, Savannah, Georgia
  - Research Facility, Arlington Heights, Illinois
  - Research Facility, Chicago, Illinois
  - Research Facility, Topeka, Kansas
  - Research Facility, Louisville, Kentucky
  - Research Facility, Baton Rouge, Louisiana
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Baltimore, Maryland
  - Research Facility, Chevy Chase, Maryland
  - Research Facility, Reisterstown, Maryland
  - Research Facility, Boston, Massachusetts
  - Research Facility, Columbia, Michigan
  - Research Facility, Minneapolis, Minnesota
  - Research Facility, Rochester, Minnesota
  - Research Facility, Tupelo, Mississippi
  - Research Facility, Kansas City, Missouri
  - Research Facility, St Louis, Missouri
  - Research Facility, Omaha, Nebraska
  - Research Facility, Scottsbluff, Nebraska
  - Research Facility, Egg Harbor, New Jersey
  - Research Facility, Binghamton, New York
  - Research Facility, Garden City, New York
  - Research Facility, Great Neck, New York
  - Research Facility, Huntington, New York
  - Research Facility, New York, New York
  - Research Facility, Rochester, New York
  - Research Facility, Troy, New York
  - Research Facility, Charlotte, North Carolina
  - Research Facility, Wilmington, North Carolina
  - Research Facility, Bismarck, North Dakota
  - Research Facility, Fargo, North Dakota
  - Research Facility, Akron, Ohio
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Dayton, Ohio
  - Research Facility, Warren, Ohio
  - Research Facility, Portland, Oregon
  - Research Facility, Beaver Falls, Pennsylvania
  - Research Facility, Philadelphia, Pennsylvania
  - Research Facility, York, Pennsylvania
  - Research Facility, Columbia, South Carolina
  - Research Facility, Kingsport, Tennessee
  - Research Facility, Memphis, Tennessee
  - Research Facility, Nashville, Tennessee
  - Research Facility, Austin, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Murray, Utah
  - Research Facility, Ogden, Utah
  - Research Facility, Burlington, Vermont
  - Research Facility, Chesapeake, Virginia
  - Research Facility, Redmond, Washington
  - Research Facility, Milwaukee, Wisconsin
- Belarus (4):
  - Research Facility, Gornel, Gormel
  - Research Facility, Hrodna, Grodnenskaya
  - Research Facility, Minsk, Minsk City
  - Research Facility, Vitebsk, Vitebsk Oblast
- Canada (14):
  - Research Facility, Edmonton, Alberta
  - Research Facility, Abbotsford, British Columbia
  - Research Facility, Vancouver, British Columbia
  - Research Facility, Guelph, Ontario
  - Research Facility, Hamilton, Ontario
  - Research Facility, London, Ontario
  - Research Facility, Ottawa, Ontario
  - Research Facility, Toronto, Ontario
  - Research Facility, Lévis, Quebec
  - Research Facility, Longheuil, Quebec
  - Research Facility, Montreal, Quebec
  - Research Facility, Québec, Quebec
  - Research Facility, Rimouski, Quebec
  - Research Facility, Saskatoon, Saskatchewan
- Croatia (2):
  - Research Facility, Zagreb, City of Zagreb
  - Research Facility, Rijeka, Rijeka
- Czechia (5):
  - Research Facility, Kralove, Kralove
  - Research Facility, Pavlov, Pavlov
  - Research Facility, Prague, Praha 2
  - Research Facility, Strakonice, Strakonice
  - Research Facility, Ústí nad Labem, Usti nad Labem
- Estonia (2):
  - Research Facility, Tallinn, Tallinn
  - Research Facility, Tartu, Tartu
- Hungary (3):
  - Research Facility, Argenti Dome Ter, Argenti Dome Ter
  - Research Facility, Budapest, Budapest
  - Research Facility, Nagyerdei Krt, Nagyerdei Krt
- Research Facility, Riga, Rīga, Latvia
- Lithuania (3):
  - Research Facility, Kaunas, Kaunas County
  - Research FacilityPanevezys, Panevezys, Panevėžys
  - Research Facility, Santariskiu, Vilnius County
- Poland (8):
  - Research Facility, Bydgoszcz, Bydgoszcz
  - Research Facility, Częstochowa, Czestochowa
  - Research Facility, Krakow, Krakow
  - Research Facility, Pruszków, Pruszkow
  - Research Facility, Sopot, Sopot
  - Research Facility, Warsaw, Warszawa
  - Research Facility, Wtoctawek, Wtoctawek
  - Research Facility, Lodz, Łódź Voivodeship
- Research Facility, San Juan, Puerto Rico
- Romania (3):
  - Research Facility, Bucharest, București
  - Research Facility, Cluj-Napoca, Cluj-napoca
  - Research Facility, Iași, Iaşi
- Russia (3):
  - Research Facility, Moscow, Mowcow
  - Research Facility, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Research Facility, Saint Petersburg, Sankt-Peterburg
- Serbia (2):
  - Research Facility, Belgrade, Beograd
  - Research Facility, Novi Sad, Novi Sad
- Ukraine (5):
  - Research Facility, Kharkiv, Kharkivs’ka Oblast’
  - Research Facility, Kyiv, Kyiv Oblast
  - Research Facility, Zabolotnogo, Odesa Oblast
  - Research Facility, Simpheropol, Simpheropol
  - Research Facility, Zaporizhzhya, Zaporizhzhya

REFERENCES:
- See also: Related Info — http://www.asacol.com/